CLINICAL TRIAL: NCT02966561
Title: Effects of a Brief Pedometer-based Behavioural Intervention for Individuals With COPD During In-patient Pulmonary Rehabilitation on 6-weeks and 6-months Objectively Measured Physical Activity - A Randomised Controlled Trial
Brief Title: Pedometer-based Behavioural Intervention for Individuals With COPD to Stay Active After Rehabilitation
Acronym: STAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg (Other)
Collaborators: Bad Reichenhall Clinic, Center for Rehabilitation, Pulmonology and Orthopedics (Unknown); German Statutory Pension Insurance (Other)
Responsible Party: Principal Investigator, Prof. Dr. Klaus Pfeifer, Prof. Dr., University of Erlangen-Nürnberg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5.011-6.031.115
Record Dates: First submitted 2016-10-07; First posted 2016-11-17 (Estimated); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Pulmonary Rehabilitation; Physical Activity; Behaviour Change; Pedometer
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity | interventions — Exercise; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pedometer-based activity promotion (Experimental): In the context of pulmonary rehabilitation (standard care), the intervention group (IG) additionally receives a pedometer-based physical activity behaviour change intervention (BCI).
  Interventions: Behavioral: Pedometer-based activity promotion; Other: Pulmonary rehabilitation (Standard care)
- Short patient education and exercise (Active Comparator): In the context of pulmonary rehabilitation (standard care), the control group (CG) additionally receives a short patient education in combination with related exercise.
  Interventions: Behavioral: Short patient education and exercise; Other: Pulmonary rehabilitation (Standard care)

INTERVENTIONS:
Behavioral: Pedometer-based activity promotion — The central components of the 2 x 45 minutes lasting pedometer-based physical activity behaviour change intervention BCI are the following behaviour change techniques (BCTs):
  * Instruction on how, where and when to perform the behaviour
  * Prompt goal setting for physical activity
  * Prompt self-monitoring of behaviour
  * Feedback on behaviour. Participants receive a pedometer and a booklet with a physical activity diary and associated information on the importance of goal setting and keeping a physical activity diary, exercise recommendations, possibilities to stay active after rehabilitation and appropriate physical activities.
  Arms: Pedometer-based activity promotion
Behavioral: Short patient education and exercise — The central components of the 2 x 45 minutes lasting intervention are revisions of knowledge of the pulmonary rehabilitation (standard care) in combination with related exercises:
  * Revision of knowledge on exercise recommendations
  * Revision of knowledge on possibilities of self-regulation of endurance training exercise intensity with the rate of perceived exertion (BORG-Scale)
  * Revision of self-regulation of endurance exercise intensity
  * Revision of strengthening activities consistent with the exercise recommendations.
  Participants receive a booklet with information on the rate of perceived exertion, exercise recommendations, possibilities to stay active after rehabilitation and appropriate physical activities.
  Arms: Short patient education and exercise
Other: Pulmonary rehabilitation (Standard care) — Standard care is an in-patient pulmonary rehabilitation (PR) in a specialized German Rehabilitation Clinic. PR is a comprehensive, multidisciplinary intervention based on a patient assessment followed by a combination of patient-tailored therapies. PR lasts on average 25 days. PR includes the following obligatory main components: Checking and, if required, adjusting the current COPD medication according to current COPD-guidelines; physical training (4-5 units/week endurance training [45 min] and 3 units/week of strength training [45 min] per week, 7 units/week whole body vibration muscle training/week); structured COPD-patient education (6 hours patient education COPD + 1 hour device training); respiratory physiotherapy in groups [2-4 units/week with 45 min]. PR is implemented by an interdisciplinary rehabilitation team.

SUMMARY:
The STAR-study (STay Active after Rehabilitation) investigates in a randomized controlled trial (RCT) the additional effect of a pedometer-based behavior change intervention (BCI) during in-patient pulmonary rehabilitation (PR) on objectively measured physical activity (PA) 6-weeks and 6-months post PR. The BCI uses the behaviour change techniques a) instruction on how, where and when to perform the behavior, b) prompt goal setting for physical activity, c) prompt self-monitoring of behavior and d) feedback on behavior. The primary outcome of PA will be measured using an accelerometer (Actigraph wGT3X) for a time period of seven days, firstly two weeks before rehabilitation begins (T0 = study phase I) as well as six weeks and six months (T3 and T4) after PR. Additionally to predict PA progression after PR, a complex personal diagnostic, including questionnaires as well as functional assessments, is to be carried out at the start (T1 = start of study phase II) and end of PR (T2). This diagnostic is based on the main ideas of the PA-related health competence model (PARC-model) and especially incorporates physical and psychological personal determinants of PA.

DETAILED DESCRIPTION:
A detailed description will be available in the study protocol publication which is generated at the moment (August, 2016).

ELIGIBILITY:
Inclusion Criteria:

* Main diagnosis for the Pulmonary Rehabilitation is an International Classification of Diseases-Code J44.- (Other chronic obstructive pulmonary disease) at all 2011 Global Initiative for Chronic Obstructive Lung Disease (GOLD) Classifications A-D and stages 1-4.

Exclusion Criteria:

* Considerably reduced health status (severe concomitant disease, which will affect the results of the outcome parameters, for example, cancer or severe cardiac, neurological or orthopaedic comorbidities)
* Considerable reduction of sight and hearing
* Severe psychiatric condition as secondary diagnosis
* Lack of ability to speak German

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 418 (Actual)
Dates: Start 2016-06; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Changes in objectively measured physical activity | 2 weeks before pulmonary rehabilitation (T0), 6 weeks after pulmonary rehabilitation (T3) and 6 months after pulmonary rehabilitation (T4)
  On each measurement occasion physical activity is going to be measured on seven consecutive days with a 3-axis accelerometer (Actigraph wGT3X-BT)

SECONDARY OUTCOMES:
Body-mass index, obstruction, dyspnea, and exercise (BODE index) | During the first week of pulmonary rehabilitation (T1); During the third and thus last week of pulmonary rehabilitation (T2)
  Questionnaire: Including body-mass index, airflow obstruction (FEV1), dyspnea (MRC-dyspnea scale) and exercise capacity (6-Min-Walk-Test)
Baseline dyspnea index (BDI) and transitional dyspnea Index (TDI) | During the first week of pulmonary rehabilitation (T1); During the third and thus last week of pulmonary rehabilitation (T2); 6 weeks after pulmonary rehabilitation (T3) and 6 months after pulmonary rehabilitation (T4)
  Questionnaire: Baseline and transitional dyspnea
Dyspnea, cough, sputum, pain | During the first week of pulmonary rehabilitation (T1); During the third and thus last week of pulmonary rehabilitation (T2); 6 weeks after pulmonary rehabilitation (T3) and 6 months after pulmonary rehabilitation (T4)
  Questionnaire: Numeric Rating Scales (self-developed)
COPD-Anxiety Questionnaire (CAF) | During the first week of pulmonary rehabilitation (T1); During the third and thus last week of pulmonary rehabilitation (T2); 6 months after pulmonary rehabilitation (T4)
  Questionnaire: COPD specific anxiety
Patient Health Questionnaire (PHQ-D9) | During the first week of pulmonary rehabilitation (T1); During the third and thus last week of pulmonary rehabilitation (T2); 6 months after pulmonary rehabilitation (T4)
  Questionnaire: Depression
St. Georges Respiratory Questionnaire (SGRQ) | 2 weeks before pulmonary rehabilitation (T0); During the first week of pulmonary rehabilitation (T1); During the third and thus last week of pulmonary rehabilitation (T2); 6 weeks (T3) and 6 months (T4) after pulmonary rehabilitation
  Questionnaire: Health-related quality of life
COPD Assessment Test (CAT) | 2 weeks before pulmonary rehabilitation (T0); During the first week of pulmonary rehabilitation (T1); During the third and thus last week of pulmonary rehabilitation (T2); 6 weeks (T3) and 6 months (T4) after pulmonary rehabilitation
  Questionnaire: Impact of COPD on health status
Control competence for physical training, physical activity-specific mood regulation and self-control, physical activity-related self efficacy, psychological need satisfaction in exercise | During the first week of pulmonary rehabilitation (T1); During the third and thus last week of pulmonary rehabilitation (T2)
  Questionnaire: Facets of physical activity-related health competence (PARC-Model)
Single-target Implicit Association Test (ST-IAT) | During the first week of pulmonary rehabilitation (T1); During the third and thus last week of pulmonary rehabilitation (T2)
  Computer-based test: Automatic affect towards physical activity
Stage of change algorithm for physical activity | During the first week of pulmonary rehabilitation (T1); During the third and thus last week of pulmonary rehabilitation (T2)
  Questionnaire: Adapted based on the transtheoretical model (TTM)
Sport- and Movement-related Self-Concordance (SSK) | During the first week of pulmonary rehabilitation (T1); During the third and thus last week of pulmonary rehabilitation (T2)
  Questionnaire: Self-concordance/ quality of motivation
Affective explicit attitudes towards performing sports activities | During the first week of pulmonary rehabilitation (T1); During the third and thus last week of pulmonary rehabilitation (T2)
  Questionnaire: Explicit cognitive and affective attitudes toward sports activities
Breathlessness Catastrophizing | During the first week of pulmonary rehabilitation (T1); During the third and thus last week of pulmonary rehabilitation (T2); 6 months after pulmonary rehabilitation (T4)
  Questionnaire: Breathlessness Catastrophizing Scale
Intolerance of Uncertainty Scale (UI-18) | During the first week of pulmonary rehabilitation (T1); During the third and thus last week of pulmonary rehabilitation (T2); 6 months after pulmonary rehabilitation (T4)
  Questionnaire: Disposition to react negative on uncertain situations
Life Orientation Test-Revised (LOT-R) | During the first week of pulmonary rehabilitation (T1); During the third and thus last week of pulmonary rehabilitation (T2); 6 months after pulmonary rehabilitation (T4)
  Questionnaire: Dispositional optimism
6 Minute Walking Test | During the first week of pulmonary rehabilitation (T1); During the third and thus last week of pulmonary rehabilitation (T2)
  Functional Test
Satisfaction with the pulmonary rehabilitation | During the third and thus last week of pulmonary rehabilitation (T2)
  Questionnaire (self-developed): Satisfaction with interventional components of the pulmonary rehabilitation
Demographic characteristics | During the first week of pulmonary rehabilitation (T1)
  Questionnaire: sex, age, height, marital status, education, weight, self-reported work status
Social medical characteristics | During the first week of pulmonary rehabilitation (T1)
  Initial physical examination including diagnosis, medication, smoking status, lung function
Sick days and use of health care services | 6 weeks after pulmonary rehabilitation (T3); 6 months after pulmonary rehabilitation (T4)
  Questionnaire: Days of incapacity to work, days in hospital, COPD-related emergency treatment
Fear avoidance COPD | During the first week of pulmonary rehabilitation (T1); During the third and thus last week of pulmonary rehabilitation (T2); 6 months after pulmonary rehabilitation (T4)
  Questionnaire: COPD disease-related fears
Self-reported physical activity | 2 weeks before pulmonary rehabilitation (T0), 6 weeks after pulmonary rehabilitation (T3) and 6 months after pulmonary rehabilitation (T4)
  Questionnaire: Physical Activity, Exercise, and Sport

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Pfeifer, Prof. Dr., Principal Investigator — Friedrich-Alexander University Erlangen-Nürnberg (FAU), Germany; Wolfgang Geidl, Dr., Principal Investigator — Friedrich-Alexander University Erlangen-Nürnberg (FAU), Germany; Konrad Schultz, Dr., Principal Investigator — Bad Reichenhall Clinic, Center for Rehabilitation, Pulmonology and Orthopedics, Bad Reichenhall, Germany
Locations (1):
- Bad Reichenhall Clinic, Center for Rehabilitation, Pulmonology and Orthopedics, Bad Reichenhall, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Geidl W, Semrau J, Streber R, Lehbert N, Wingart S, Tallner A, Wittmann M, Wagner R, Schultz K, Pfeifer K. Effects of a brief, pedometer-based behavioral intervention for individuals with COPD during inpatient pulmonary rehabilitation on 6-week and 6-month objectively measured physical activity: study protocol for a randomized controlled trial. Trials. 2017 Aug 29;18(1):396. doi: 10.1186/s13063-017-2124-z. PMID 28851462
- [Result] Geidl W, Carl J, Cassar S, Lehbert N, Mino E, Wittmann M, Wagner R, Schultz K, Pfeifer K. Physical Activity and Sedentary Behaviour Patterns in 326 Persons with COPD before Starting a Pulmonary Rehabilitation: A Cluster Analysis. J Clin Med. 2019 Aug 29;8(9):1346. doi: 10.3390/jcm8091346. PMID 31470678
- [Result] Janssens T, Van de Moortel Z, Geidl W, Carl J, Pfeifer K, Lehbert N, Wittmann M, Schultz K, von Leupoldt A. Impact of Disease-Specific Fears on Pulmonary Rehabilitation Trajectories in Patients with COPD. J Clin Med. 2019 Sep 13;8(9):1460. doi: 10.3390/jcm8091460. PMID 31540306
- [Derived] Carl J, Schultz K, Janssens T, von Leupoldt A, Pfeifer K, Geidl W. The "can do, do do" concept in individuals with chronic obstructive pulmonary disease: an exploration of psychological mechanisms. Respir Res. 2021 Oct 6;22(1):260. doi: 10.1186/s12931-021-01854-1. PMID 34615520